CLINICAL TRIAL: NCT03192319
Title: Comparison of Change in Humoral and Cellular Immunity Induced by Zoster Vaccine According to the Timing of Vaccination After Hematopoietic Stem Cell Transplantation
Brief Title: Optimal Timing of Zoster Vaccine After Hematopoietic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Wan Beom Park, Associate Professor, Seoul National University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H1705030852
Record Dates: First submitted 2017-06-16; First posted 2017-06-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Herpes Zoster
Keywords: Herpes zoster vaccine; Cell-mediated immunity; hematopoietic stem cell transplantation
MeSH Terms: conditions — Herpes Zoster | interventions — Herpes Zoster Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 2years to 5years after HCT (Experimental): Patients will be vaccinated with Zostavax from 2years to 5years after hematopoietic stem cell transplantation
  Interventions: Biological: Zostavax
- 5years to 10years after HCT (Active Comparator): Patients will be vaccinated with Zostavax from 5years to 10years after hematopoietic stem cell transplantation
  Interventions: Biological: Zostavax
- 6 month after chemotherapy for leukemia (Active Comparator): Patients will be vaccinated with Zostavax 6 months after the leukemia is cured with chemotherapy
  Interventions: Biological: Zostavax
- healthy people (Active Comparator): Healthy adults over 50 years old will be vaccinated with Zostavax
  Interventions: Biological: Zostavax

INTERVENTIONS:
Biological: Zostavax — Zostavax will be administrated by subcutaneous injection

SUMMARY:
The purpose of this study is to determine the optimal timing of zoster vaccination to induce both higher cell-mediated immunity and humoral immunity in adult patient aged over 50 with history of hematopoietic stem cell transplantation(HSCT).

DETAILED DESCRIPTION:
Due to lack of data on safety of live vaccine in the recipient of hematopoietic stem cell transplantation, CIBMTR(Center for International Blood and Marrow Transplant Research) guidelines recommend varicella vaccination only in patients who is at least two years after transplantation and without graft versus host disease and no immunosuppressive drug.

However, recent studies have demonstrated the safety and efficacy of shingles vaccination in patients receiving hematopoietic stem cell transplantation.

But, there is no basis for timing of live vaccine administration after HSCT.

The investigators plan to make scientific recommendation for optimal timing of zoster vaccine after HSCT by comparing immune response between two groups(vaccination at 2 to 5years after HSCT vs. 5 to 10years after HSCT). Primary outcome is interferon gamma releasing ELISPOT response at week 6 after vaccination. Secondary outcome is ELISA titer for zoster-specific IgG at week 6 after vaccination.

All the patients will be asked if they have any contraindication for zoster vaccine by a physician before vaccination. And they will be monitored for any adverse reaction of the vaccination after 6 weeks(visiting the hospital).

In order to confirm the efficacy of the experiment, 30 healthy controls and 30 patients who were treated with chemotherapy alone for leukemia were selected. The control group will also apply the same protocol as above.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 50 years or older who is at least 2 years after hematopoietic stem cell transplantation (Experimental group)
* Adults aged 50 years or older who is at least 6 months after being cured by chemotherapy for leukemia (Control group)
* Healthy Adults aged 50 years or older who do not meet exclusion criteria (Control group)
* Adults who can understand and agreed with the informed consents

Exclusion Criteria:

* Adults who have conditions which is contraindication for zoster vaccine
* Adults who take immunosuppressant
* Adults with graft versus host disease(GVHD)
* Adults who take antivirals agent
* Adults who experienced VZV infection after hematopoietic stem cell transplantation
* Adults who received VZV vaccination already after hematopoietic stem cell transplantation
* Adults who are not eligible for zoster vaccination by investigator's assessment

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-08-23 (Actual); Study Completion 2018-08-23 (Actual)

PRIMARY OUTCOMES:
Varicella-zoster virus-specific interferon-gamma ELISPOT response | before Zostavax vaccination and at week 6 after vaccination
  Investigators measure the number of SFC(spot forming cells) using interferon-gamma ELISPOT(enzyme-linked immunospot) assay at both right before vaccination and week 6 after vaccination and see the change between two values.

SECONDARY OUTCOMES:
Antibody titer against varicella-zoster virus | before Zostavax vaccination and at week 6 after vaccination
  Investigators measure the titer of Varicella zoster virus (VZV)-specific Ab by enzyme-linked immunosorbent assay at both right before vaccination and week 6 after vaccination and see the fold change between two values

CONTACTS AND LOCATIONS:
Overall Officials: Park Wan Beom, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tomblyn M, Chiller T, Einsele H, Gress R, Sepkowitz K, Storek J, Wingard JR, Young JA, Boeckh MJ; Center for International Blood and Marrow Research; National Marrow Donor program; European Blood and MarrowTransplant Group; American Society of Blood and Marrow Transplantation; Canadian Blood and Marrow Transplant Group; Infectious Diseases Society of America; Society for Healthcare Epidemiology of America; Association of Medical Microbiology and Infectious Disease Canada; Centers for Disease Control and Prevention. Guidelines for preventing infectious complications among hematopoietic cell transplantation recipients: a global perspective. Biol Blood Marrow Transplant. 2009 Oct;15(10):1143-238. doi: 10.1016/j.bbmt.2009.06.019. No abstract available. PMID 19747629
- [Background] Issa NC, Marty FM, Leblebjian H, Galar A, Shea MM, Antin JH, Soiffer RJ, Baden LR. Live attenuated varicella-zoster vaccine in hematopoietic stem cell transplantation recipients. Biol Blood Marrow Transplant. 2014 Feb;20(2):285-7. doi: 10.1016/j.bbmt.2013.11.013. Epub 2013 Nov 22. PMID 24269706
- [Background] Gilbert PB, Gabriel EE, Miao X, Li X, Su SC, Parrino J, Chan IS. Fold rise in antibody titers by measured by glycoprotein-based enzyme-linked immunosorbent assay is an excellent correlate of protection for a herpes zoster vaccine, demonstrated via the vaccine efficacy curve. J Infect Dis. 2014 Nov 15;210(10):1573-81. doi: 10.1093/infdis/jiu279. Epub 2014 May 13. PMID 24823623
- [Background] Kim JW, Min CK, Mun YC, Park Y, Kim BS, Nam SH, Koh Y, Kwon JH, Choe PG, Park WB, Kim I. Varicella-zoster virus-specific cell-mediated immunity and herpes zoster development in multiple myeloma patients receiving bortezomib- or thalidomide-based chemotherapy. J Clin Virol. 2015 Dec;73:64-69. doi: 10.1016/j.jcv.2015.10.018. Epub 2015 Oct 24. PMID 26546878
- [Background] Levin MJ, Oxman MN, Zhang JH, Johnson GR, Stanley H, Hayward AR, Caulfield MJ, Irwin MR, Smith JG, Clair J, Chan IS, Williams H, Harbecke R, Marchese R, Straus SE, Gershon A, Weinberg A; Veterans Affairs Cooperative Studies Program Shingles Prevention Study Investigators. Varicella-zoster virus-specific immune responses in elderly recipients of a herpes zoster vaccine. J Infect Dis. 2008 Mar 15;197(6):825-35. doi: 10.1086/528696. PMID 18419349